CLINICAL TRIAL: NCT05840484
Title: Comprehensive Monitoring of Men With Prostate Cancer Cared for by "Active Surveillance
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-0297; NCI-2023-03146 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2023-04-11; First posted 2023-05-03 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cohort-1: Participants with localized very low- or low-risk prostate cancer meeting consensus criteria for active surveillance
  Interventions: Other: Active Surveillance
- Cohort-2: Participants with NCCN intermediate-risk localized prostate cancer requesting active surveillance (per patient and clinician shared decision making);
  Interventions: Other: Active Surveillance
- Cohort-3: Participants with severe medical comorbidities (defined as CCI estimated 10-year survival < 50% and agreed by treating clinician) and high- or very high-risk group localized prostate cancer.
  Clinical trial investigators and staff will make every effort to integrate study visits with the subjects' clinic visits during participation.
  Interventions: Other: Active Surveillance

INTERVENTIONS:
Other: Active Surveillance — Participants will be asked to complete questionnaires, have physical and rectal examinations, have prostate biopsies, and have imaging scans (such as MRIs). These visits will be done between every 6 months and every 2-3 years, depending on the test/procedure.

SUMMARY:
Prostate cancer is the most commonly diagnosed cancer in men. However, there is a wide range in prognosis determined by a host of factors. This study will evaluate the feasibility of guiding therapeutic intervention electronically facilitated symptom and disease monitoring in patients being followed on Active Surveillance. Additionally, we will develop a tissue and data resource to support discovery and hypothesis generation to evaluate germline and/or somatic alterations in relation to cancer-specific and overall outcomes..

DETAILED DESCRIPTION:
Primary objectives:

1. Monitor cancer-specific outcomes of men who meet consensus criteria for active surveillance under one of three categories: 1) low or very low-risk prostate cancer, 2) intermediate risk with patient consent, or 3) severe medical comorbidities and high-risk localized prostate cancer or patient desire, despite recommendation

Secondary objectives:

1. Screen for a relationship between cancer-specific and clinical outcomes related to selected comorbidities.
2. Determine the feasibility of electronically facilitated symptoms and disease monitoring to guide therapeutic intervention and prompt therapeutic course correction.
3. Develop a tissue and data resource to support discovery and hypothesis generation focused on germline alterations, somatic alterations, and/or the interaction between the two in determining cancer-specific and overall outcomes

ELIGIBILITY:
Inclusion criteria:

1. Patients will have histologic diagnosis of adenocarcinoma of the prostate within 24 months of study entry.
2. Patient must meet at least one of the following clinical indications for AS: National Comprehensive Cancer Network (NCCN) very low risk or low risk prostate cancer meeting consensus guidelines for AS; NCCN intermediate-risk prostate cancer requesting AS (per patient and clinician shared decision making); or have severe medical comorbidities (defined as CCI estimated 10-year survival < 50% and agreed by treating clinician) with high- or very high-risk localized prostate cancer.
3. Patients must agree to comply with the surveillance schedule.
4. Patients must be over 18 years of age
5. Written informed consent
6. Patients must be fluent in the English language to participate in the patient report outcome and symptoms monitoring portion of the trial.

Exclusion criteria:

1. Patients are ineligible if they choose not to share their medical data for research purposes.
2. Prior radiation therapy for treatment of the primary tumor.
3. Planned concomitant hormonal therapy, chemotherapy, or radiation therapy while on protocol

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: M D Anderson Cancer Center
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-03-29 (Actual); Primary Completion 2029-07-30 (Estimated); Study Completion 2029-07-30 (Estimated)

PRIMARY OUTCOMES:
To estimate the 5-year disease progression rate of patients with low or very low-risk prostate cancer who choose to undergo active surveillance with remote monitoring | through study completion; an average of 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Logothetis, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org